CLINICAL TRIAL: NCT00568984
Title: Efficacy and Safety of Repaglinide and Metformin Combined in Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Repaglinide and Metformin Combined in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-3017
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repaglinide
Drug: metformin
Drug: glicazide

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the efficacy of blood glucose control with combination therapy of repaglinide and metformin compared to conventional treatment with a sulphonylurea or metformin in monotherapy in type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months
* No previous treatment for diabetes
* HbA1c between 7.0-12.0%
* Body Mass Index (BMI) between 19.0-40.0 kg/m2

Exclusion Criteria:

* Type 1 diabetes
* Known unstable/untreated proliferative retinopathy
* Uncontrolled treated/untreated hypertension
* Pregnancy, breast-feeding, the intention of becoming pregnant or judged to be using inadequate contraceptive measures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2002-11-21 (Actual); Primary Completion 2003-11-10 (Actual); Study Completion 2003-11-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 16 weeks of treatment

SECONDARY OUTCOMES:
Glucose profiles
Quality of life assessment
Treatment satisfaction
Hypoglycaemic events
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- China (2):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Ipoh
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
- Philippines (6):
  - Novo Nordisk Investigational Site, Cebu City
  - Novo Nordisk Investigational Site, Manila
  - Novo Nordisk Investigational Site, Marikina City
  - Novo Nordisk Investigational Site, Pampanga
  - Novo Nordisk Investigational Site, Quezon
  - Novo Nordisk Investigational Site, Quezon City
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com